CLINICAL TRIAL: NCT03539757
Title: Development of Novel MRI Methods for Detecting, Discriminating, and Measuring Liver Fibrosis and Congestion in Fontan Patients
Status: Terminated | Type: Observational
Why Stopped: Due to lack of enrollment this study was permanatly closed March 2022. The incidence of FONTAN patients being referred for liver biospsies and occurance of COVID effected participants enrolled.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_FALD MRI
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2021-06

CONDITIONS: Liver Fibrosis
Keywords: Liver fibrosis; Fontan surgery; MRI; Novel Methods
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Fontan patients: Pediatric and adult Fontan patients will undergo MRI (Magnetic Resonance Imaging) of the liver using novel, non-contrast MRI methods. These MR methods will be used to detect, discriminate and measure liver fibrosis and congestion. The resulting quantitative imaging measurements will be correlated with histopathologic data obtained from a clinically-indicated liver biopsy.
  Interventions: Device: Non-Contrast Magnetic Resonance Imaging

INTERVENTIONS:
Device: Non-Contrast Magnetic Resonance Imaging — The investigators plan to prospectively assess the correlation of liver fibrosis and congestion measurements obtained from novel, non-contrast MR imaging methods to histopathologic data obtained from a clinically-indicated liver biopsy in Fontan patients.

SUMMARY:
In this research study, the investigators will conduct a prospective cross-sectional study of pediatric and adult Fontan patients that will correlate a variety of quantitative MRI biomarkers with histopathologic data.

DETAILED DESCRIPTION:
The purpose of this study is to develop noninvasive MRI methods for detecting, discriminating, and measuring liver fibrosis and congestion in the adolescent and adult Fontan population by correlating quantitative imaging measurements with histopathologic data, using a cross-sectional approach.

Over 5 years, approximately 40 pediatric and adult subjects (approximately 8 subjects per year) undergoing clinically-indicated liver biopsy for the evaluation of either 1) focal liver lesions/masses, or 2) suspected liver fibrosis/parenchymal disease will be recruited to participate in this study. Subjects will undergo research MR imaging within ±2 weeks of the liver biopsy procedure. A variety of MRI biomarkers will be correlated with histopathologic data obtained from the clinically indicated liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Single ventricle physiology congenital heart disease status post Fontan palliation
* Undergoing clinically-indicated liver biopsy
* Ability to tolerate 60 minutes in an MRI scanner without sedation

Exclusion Criteria:

* Known contraindication to MR imaging (e.g., implanted non-MRI compatible device)
* Known or suspected pregnancy. Female subjects of child bearing potential will undergo urine pregnancy testing prior to imaging

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects will be identified through Cincinnati Children's Hospital Medical Center's (CCHMC) cardiology or hepatology clinics, or through CCHMCs Fontan Management Program
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
MR elastography data correlation to histologic data | 60 minutes
  MR elastography of the liver data will be correlated with histopathologic data obtained from non-lesional liver tissue. Histologic fibrosis and congestion will be scored by a pathologist using semi-quantitative grading systems (e.g., METAVIR scoring system for fibrosis

SECONDARY OUTCOMES:
MR T1 mapping data (corrected and uncorrected) correlation to histologic data | 60 minutes
  MR T1 mapping liver data (corrected and uncorrected) will be correlated with histopathologic data obtained from non-lesional liver tissue. Histologic fibrosis and congestion will be scored by a pathologist using semi-quantitative grading systems (e.g., METAVIR scoring system for fibrosis)
MR T1rho data correlation to histologic data | 60 minutes
  MR T1rho liver data will be correlated with histopathologic data obtained from non-lesional liver tissue. Histologic fibrosis and congestion will be scored by a pathologist using semi-quantitative grading systems (e.g., METAVIR scoring system for fibrosis)
MR T2 mapping data correlation to histologic data | 60 minutes
  MR T2 mapping liver data will be correlated with histopathologic data obtained from non-lesional liver tissue. Histologic fibrosis and congestion will be scored by a pathologist using semi-quantitative grading systems (e.g., METAVIR scoring system for fibrosis)
MR Diffusion weighted data correlation to histologic data | 60 minutes
  MR Diffusion weighted liver data will be correlated with histopathologic data obtained from non-lesional liver tissue. Histologic fibrosis and congestion will be scored by a pathologist using semi-quantitative grading systems (e.g., METAVIR scoring system for fibrosis)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, MD,MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No